CLINICAL TRIAL: NCT06689397
Title: Investigating Epstein-Barr Virus Associated Conjunctivitis
Acronym: EBV Conj
Status: Enrolling by invitation | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: LARF1028; 342525 (Other: IRAS); 24/YH/0160 (Other: Research Ethics Committee)
Record Dates: First submitted 2024-09-08; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Conjunctivitis; EBV Infection
MeSH Terms: conditions — Conjunctivitis; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Conjunctivitis means inflammation of the conjunctiva, the thin transparent layer over the white of the eye and under the eyelids. Acute conjunctivitis caused by infection is the most common condition seen in ophthalmic emergency departments, accounting for up to 10% of cases. It is responsible for 41% of eye-related general practice consultations. A diagnosis is usually made on the patient's symptoms and signs, despite this being less reliable than laboratory testing. When a cause is found, it is usually a common cold virus called adenovirus, that gets better with time and does not require treatment.

Through investigating cases of conjunctivitis at Moorfields, it has been discovered that in addition to adenovirus, Epstein Barr virus (EBV) is sometimes detected in conjunctival swabs from individuals with conjunctivitis. EBV is a very common viral infection that 95% of adults have experienced. EBV infection mostly passes unnoticed but when symptoms do occur, they include a sore throat, high temperature, swollen glands and tiredness, often called glandular fever or infectious mononucleosis. Conjunctivitis can also occur. EBV remains in the body after infection and rarely causes further problems. The virus can become active again occasionally, which is known as reactivation.

Reactivation usually passes unnoticed but sometimes is associated with recurrence of symptoms. It is possible that reactivation may cause conjunctivitis. It is not certain, which is will be observed as a part of this study, as it might be the cause of some of the conjunctivitis seen.

Through a collaboration with University College London (UCL), the aim is to gain further insight into infectious conjunctivitis, particularly in relation to EBV. This will be done by taking a swab of the conjunctiva, a single blood test and a tiny (1-2mm) tissue sample from the inner eyelid. Improved knowledge will allow the research team to develop better guidance and treatment for patients with conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Participants shall be considered eligible for inclusion if:

  * Aged ≥16 years;
  * working diagnosis of infective (viral) follicular conjunctivitis (<4 weeks duration)
  * EBV positive conjunctival swab

Exclusion Criteria:

* • Present with symptoms/signs such that another diagnosis is deemed more likely, for example topical medication-induced conjunctivitis.

  * Participant declines diagnostic tests or appropriate corneal or conjunctival sample(s) not obtained for any reason

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from Moorfields A&E. Eligible patients will be identified by a member of the clinical triage team. All eligible patients will be enrolled during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
The number of participants with clinically suspected viral conjunctivitis in which EBV DNA is identified on NAAT. | From enrollment to the end of visit 2 which can occur within up to 7 days from enrollment.
  To confirm the proportion of:
  * participants with clinically suspected viral conjunctivitis in which EBV DNA is identified on NAAT.
  * EBV NAAT-positive participants who have a new EBV infection versus those with a reactivation of earlier disease.
  * participants in whom EBV is confirmed the cause of conjunctivitis on further investigation.

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No